CLINICAL TRIAL: NCT06482684
Title: Early Treatment Intensification in Patients With High Risk Mantle Cell Lymphoma Using CAR-T-cell Treatment After an Abbreviated Induction Therapy With Rituximab and Ibrutinib and 6 Months Ibrutinib Maintenance (Arm A) as Compared to Standard of Care Induction and Maintenance (Arm B)
Brief Title: CAR-T-cell Treatment for Untreated High Risk MANtle Cell Lymphoma
Acronym: CARMAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christian Schmidt, MD (Other)
Collaborators: Johannes Gutenberg University Mainz (Other)
Responsible Party: Sponsor-Investigator, Christian Schmidt, MD, Head of Study Center, Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARMAN; 2022-502405-15-01 (EU CTIS Number)
Record Dates: First submitted 2024-06-26; First posted 2024-07-01 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Mantle Cell Lymphoma
Keywords: High Risk MCL; CAR-T-Cells; MCL Firstline Treatment
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — brexucabtagene autoleucel; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm A (Experimental): The abbreviated induction phase consists of 2 cycles of Ibrutinib + Rituximab and 2 cycles of Ibrutinib + R-CHOP for primary tumor reduction followed by CAR-T-cell treatment. In case of good clinical response (PR or CR) after 2 cycles of Ibrutinib + Rituximab, Ibrutinib + R-CHOP can be omitted. In this case, one cycle of Ibrutinib monotherapy will be applied. T cell apheresis will be performed after the initial 2 cycles. Application of KTE-X19 will be performed after lymphodepleting chemotherapy with Fludarabine and Cyclophosphamide (FC). After stable hematopoietic recovery, maintenance with Ibrutinib will be applied for 6 months but not prior to day 60 post CAR. The follow-up period starts after the completion of Ibrutinib maintenance and takes 4.5 up to 7 years.
  Interventions: Drug: KTE-X19; Drug: Ibrutinib
- Arm B (Active Comparator): Younger patients (≤ 65 years) will receive 3 cycles R-CHOP + Ibrutinib/ 3 cycles R-DHAP alternating, followed by autologous stem cell transplantation (ASCT). Elderly patients (≥ 65 years) will receive 6 cycles of Bendamustine and Rituximab + Ibrutinib or R-CHOP + Ibrutinib without ASCT. Independently of age, control patients receive 2 years of maintenance therapy with Ibrutinib and 3 years of Rituximab maintenance if foreseen by national guidelines, in addition to Ibrutinib maintenance.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: KTE-X19 — See description of treatment arms
  Arms: Arm A
Drug: Ibrutinib — See description of treatment arms

SUMMARY:
First-line CAR-T-cell consolidation after an abbreviated induction with 2 cycles of Rituximab and Ibrutinib prior to CAR-T-cell treatment and followed by 6 months of maintenance with Ibrutinib in patients with high risk MCL.

DETAILED DESCRIPTION:
This phase II clinical trial will compare the efficacy, safety and tolerability of first-line treatment with KTE-X19 after a shortened induction with Rituximab and Ibrutinib to conventional immunochemotherapy and Ibrutinib followed by ASCT in younger patients in high-risk MCL patients or immunochemotherapy plus BTKi for elderly, but still fit patients (need to be CAR-T-cell eligible). As primarily the potential of CAR-T-cell treatment is evaluated within this trial, in case of failure to achieve a partial response will be treated with 2 additional cycles of R-CHOP, which can be omitted in case of sufficient response to Ibrutinib-based treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of MCL according to WHO classification, with documentation of either overexpression of cyclin D1 or presence of t(11;14)
2. At least one High Risk MCL - feature as defined as I. MIPI-c high intermediate (HI) or high (H) risk (i.e. high risk MIPI irrespective of Ki-67 or intermediate risk MIPI and Ki-67>=30% (Ki-67 based on local pathology) and/or II. TP53-mutation and/or TP53-overexpression by immunohistochemistry (> 50% of lymphoma cells)
3. No prior treatment for MCL
4. Stage II-IV (Ann Arbor)
5. 18-75 years
6. At least 1 measurable lesion according to the Lugano Response Criteria (>1.5 cm nodal lesion or > 1cm extranodal lesion); in case of bone marrow infiltration only, bone marrow aspiration and biopsy is mandatory for all staging evaluations.
7. ECOG performance status ≤ 2
8. The following laboratory values at screening (unless discrepancies are related to MCL):

   I. Absolute neutrophil count (ANC) ≥ 1000 cells/μL II. Platelets ≥75,000 cells/μL III. Creatinine <2 mg/dL or calculated creatinine clearance ≥60 mL/min IV. Transaminases (AST and ALT) < 2.5 x ULN V. Total bilirubin <= 2 x ULN unless other reason known (e.g. Gilbert-Meulengracht-Syndrome, or due to lymphoma involvement)
9. No evidence of CNS-disease
10. Written informed consent form according to ICH/EU GCP and national regulations, ability to follow study instructions and likely to attend and complete all required visits
11. Sexually active men and women of child-bearing potential must agree to use one of the highly effective contraceptive methods (combined oral contraceptives using two hormones, contraceptive implants, injectables, intrauterine devices, sterilized partner) together with one of the barrier methods (latex condoms, diaphragms, contraceptive caps) while on study; this should be maintained for 6 months after the last dose of KTE-X19 or for 3 months after last dose of Ibrutinib, whichever is longer
12. Negative serum or urine pregnancy test (Females of childbearing potential only, Females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential)
13. Willingness not to drive a motor vehicle for 8 weeks post CAR T cell treatment
14. Possibility to reach the site within 2 hours in case of toxicity / emergency

Exclusion Criteria:

1. Subjects not able to give consent
2. Subjects without legal capacity, unable to understand the nature, scope, significance and consequences of this clinical study
3. Known history of hypersensitivity to the investigational drug, to drugs with a similar chemical structure or to aminoglycosides
4. Simultaneously active participation in another clinical study involving an investigational medicinal product within 30 days prior to enrollment. Patients included in follow up periods of other clinical trials without ongoing trial medication are allowed
5. Subjects with a physical or psychiatric condition which at the investigator's discretion may put the subject at risk, may confound the study results, or may interfere with the subject's participation in this clinical study
6. Known or persistent abuse of medication, drugs or alcohol
7. Serious concomitant disease interfering with a regular therapy according to the study protocol:

   I. Clinically significant cardiovascular disease such as symptomatic arrhythmias, congestive heart failure, higher grade AV-block, unstable angina, myocardial infarction, cardiac angioplasty or stenting within 12 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification or LVEF below 50% II. Baseline oxygen saturation ≤ 92% on room air III. Clinical significant pleural effusion (if not lymphoma related) IV. Endocrinological (severe, not sufficiently controlled diabetes mellitus)
8. Current or planned pregnancy or nursing women. History of or active malignancy other than MCL, non-melanoma skin cancer, carcinoma in situ (e.g. cervix, bladder, breast) or prostate cancer unless disease-free for at least 3 years (and PSA within normal range in case of prostate cancer).
9. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management.
10. Positive test results for chronic HBV infection (defined as positive HBsAg serology) (mandatory testing) Patients with occult or prior HBV infection (defined as negative HBsAg and positive total HBcAb) may be included if HBV DNA is undetectable
11. Positive test results for hepatitis C (mandatory hepatitis C virus [HCV] antibody serology testing). Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA
12. Patients with known HIV infection (mandatory test)
13. History or presence of CNS disorder, such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, cerebral edema, posterior reversible encephalopathy syndrome, or any autoimmune disease with CNS involvement
14. History of or active autoimmune disease (e.g. Crohn's disease, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression / systemic medication within the last 2 years
15. History of deep vein thrombosis or pulmonary embolism requiring therapeutic anticoagulation within 6 months of enrolment
16. Known severe primary immunodeficiency
17. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment
18. Live vaccine ≤ 6 weeks prior to planned start of study treatment
19. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow up schedule

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2031-06-15 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure Free Survival | From Randomization to any to any discontinuation of the per protocol treatment due to stable or progressive disease
  Time from randomization to any discontinuation of the per protocol treatment due to stable or progressive disease during induction, stable disease at the end of induction, progressive disease at any time after end of induction treatment and death from any cause, whichever occurred first. Stable disease at end of induction is defined as failure event because it represents a regular indication for salvage treatment in MCL.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | from the date of response (CR or PR within 6 months from randomization) to progression or death from any cause
Complete remission (CR) rate | 6 months from randomization until end of trial
Time to first response | date of randomization to the date of first response (CR or PR)
Overall survival | day 1 after randomization until end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Georg Hess, MD, Principal Investigator — Johannes Gutenberg University Mainz
Locations (2):
- Germany (2):
  - University Hospital of Mainz, Mainz
  - Klinikum der Universität München, Munich

REFERENCES:
- [Derived] Silkenstedt E, Dreyling M. First Line Therapy in Mantle Cell Lymphoma-The Role of BTKi in the Initial Treatment of Transplant-Eligible and -Ineligible Patients. Hematol Oncol. 2025 Jun;43 Suppl 2(Suppl 2):e70073. doi: 10.1002/hon.70073. PMID 40517546